CLINICAL TRIAL: NCT04565041
Title: Can Social Support Figures Enhance Fear Extinction in Patients With Social Anxiety?
Brief Title: Social Support and Enhanced Fear Extinction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SSE; R21MH125274 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Fear; Anxiety
Keywords: social support; fear extinction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Social Support (Experimental)
  Interventions: Behavioral: Social Support

INTERVENTIONS:
Behavioral: Social Support — Presence of an image of a social support figure (provided by participant) during a fear extinction procedure

SUMMARY:
University of California, Los Angeles researchers will recruit healthy participants and anxious participants (those diagnosed with social anxiety disorder) age 18-55 years old to participate in a study examining whether the ability of social support figure reminders to enhance the extinction of fear in healthy participants extends to those with anxiety disorders.

After being recruited from the UCLA community (healthy participants, n = 50) or referred by treatment providers at the Anxiety and Depression Research Center at UCLA (anxious participants, n = 50) and undergoing a telephone screening and in-person screening, 100 participants will be enrolled in the study, with an expected recruited 150 to reach this number. During the experiment, all participants will undergo the same procedures: undergoing a fear extinction procedure in which threatening cues--cues that predict electric shock--will be paired with either an image of a social support figure (provided by participants) or an image of a smiling stranger. These pairings will be presented repeatedly in the absence of shock in order for fear extinction to occur. Participants will return for a follow-up test to determine if fear extinction was successful.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 18 to 55
* fluent in English
* no history of mental illness (healthy participants: including anxiety, depression, phobia, or any other mental health related disorder diagnosed by a mental health professional)
* diagnosis of social anxiety disorder (anxious participants: allowed co-morbid disorders include depression, other anxiety disorders, and PTSD)

Exclusion Criteria:

* pregnant or planning to become pregnant during the experiment period
* presence of chronic mental illness (healthy participants: as determined by the report of a past diagnosis of mental illness by a physician or psychologist and/or the prescription of medication related to mental health disorder; including anxiety, depression, phobia, or any other diagnosed psychological disorder)
* presence of non-allowed co-morbid disorders (anxious participants: including, bipolar disorder, psychosis, substance use disorder, neurological disorder, and/or obsessive-compulsive disorder)
* current and regular use of prescription medications related to mental health disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Fear response directly post-extinction | within experimental session - directly post-extinction procedure
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).
Fear response 24 hours post-extinction | 24 hours following the completion of fear extinction procedures
  presence of fear response as indicated by significantly higher galvanic skin response (GSR: an index of peripheral stress responding) to a previously learned fearful image (CS+) compared to a baseline comparator (CS-: never learned to be fearful).

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No